CLINICAL TRIAL: NCT03985111
Title: In High Risk Patients Undergoing Elective Colorectal Resection, Does Routine Placement of a Central Venous Catheter Reduce Peri-operative Fluid Administration in Theatre and the Critical Care Unit?
Brief Title: Does a Central Venous Line Reduce Perioperative Fluid Administration?
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 012593; 19/LO/0099 (Other: HREC); 252375 (Other: IRAS)
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Disorders
Keywords: perioperative care; perioperative blood pressure management; perioperative fluid management
MeSH Terms: interventions — Central Venous Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No CVC inserted: Patients undergoing major elective colorectal resection without central venous catheter inserted pre-operatively
- CVC inserted: Patients undergoing major elective colorectal resection with a central venous catheter inserted pre-operatively
  Interventions: Device: Central Venous Catheter

INTERVENTIONS:
Device: Central Venous Catheter — Insertion of a central venous catheter insertion pre-operatively (electively)
  Groups: CVC inserted

SUMMARY:
'Hypothesis-generating' study to assess whether the presence of a central venous line significantly affects the volumes of fluid infused perioperatively in major elective colorectal surgery

DETAILED DESCRIPTION:
There are several indications for elective central venous cannulation in major colorectal surgery, particularly in those at a higher risk of morbidity and mortality. These include: the ability to infuse certain vasoactive medications, monitor central venous pressure, allow for frequent blood sampling, and provide a route of access for total parenteral nutrition(1). Furthermore, there has been a great deal of recent interest in whether there are improved outcomes with restrictive as opposed to liberal fluid therapy in major abdominal surgery(2), and, similarly, with individualised, rather than generic, blood pressure management in major surgery(3). However, there have been no major studies to date examining whether the simple act of electively inserting a central venous catheter prior to the start of surgery influences the volume of fluid infused and the use of vasopressors perioperatively.

The RELIEF trial reported that modestly liberal perioperative fluid regimens conferred no greater disability-free survival benefit over restrictive regimens, but are likely to reduce rates of acute kidney injury(2). This contrasts with the restrictive protocols championed by various Enhanced Recovery After Surgery (ERAS) programs(4). Previous works have suggested that not only does adherence to ERAS principles lead to superior patient outcomes, but some have gone further in identifying restriction of intravenous fluids perioperatively to be one of the few interventions that independently predicts a better outcome(5). One of the advantages of central venous catheterisation is the ability to administer drugs in smaller volumes of fluid. Therefore, given the intensity of the debate surrounding restrictive and liberal regimens, it should be investigated whether the availability of central venous access impacts upon the volumes of fluid infused.

Furthermore, central venous catheterisation is unlikely just to have an impact via the avoidance of inadvertent larger volume infusion, which is sometimes seen with drug administration through a peripheral line. The RELIEF trial reported that the patient cohort managed with a restrictive fluid regimen were more likely to receive vasopressor support, compared with those receiving a liberal regimen(2). The presence of a central venous catheter enables the use of potent vasopressor agents, such as noradrenaline, which will further influence fluid administration, by introducing a second therapeutic option for correcting perioperative hypotension. The importance of 'tight' blood pressure control has been demonstrated by the INPRESS trial, which showed a reduction in post-operative organ dysfunction with individualised blood pressure management, over standard management strategies(3). This is of particular importance, as evidence has shown that cardiac output-directed fluid therapy should not lead to 'excessive fluid administration, but may lead to a more individualised approach to achieving the correct dose of fluid'(6), and may require concomitant use of vasoactive agents.

Thus, the investigators have set out to investigate whether the elective insertion of a central venous catheter prior to the start of major colorectal surgery, influences the volumes, and types, of fluid infused, as well as the use and mean dose of vasopressor agents, intra-operatively and for the first 12 hours post-operatively.

1. Smith, RN, et al., 'Central venous catheters', BMJ 2013; 347:f6570
2. Myles, PS, et al., 'Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery', N Engl J Med 2018; 378:24
3. Futier, E, et al., 'Effect of Individualised vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery', JAMA 2017; 318(14):1346
4. Feldheiser, A, et al., 'Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice', Acta Anaesthesiologica Scandinavia 2016, 60:289
5. Gustafsson, UO, et al., 'Adherence to the Enhanced Recovery After Surgery Protocol and Outcomes After Colorectal Cancer Surgery', Arch Surg 2011; 146(5):571
6. Pearse, RM, et al., 'Effect of a Perioperative Cardiac Output- Guided Haemodynamic Therapy Algorithm on Outcomes Following Major Gastrointestinal Surgery', JAMA 2014; 311(21):2181

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be all adult patients presenting for elective major colorectal surgery (resection), whom are to be electively admitted to critical care directly from theatre.

Exclusion Criteria:

* Patients under 18 years of age
* Patients undergoing emergency surgery
* Those not admitted electively to critical care directly from theatre
* Those patients that do not undergo any bowel resection
* Patients in whom central venous catheter insertion is as an emergency peri- operatively
* Patients refusing/unable to give valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, undergoing elective major colorectal resection, at a district general hospital in east London, UK.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Volume of intravenous fluid infused intra-operatively | Intra-operatively (from induction to leaving theatre)
  To assess whether the presence of a central venous catheter influences the volume of intravenous fluid infused intra-operatively
Volume of intravenous fluid infused post-operatively | The first 12 hours post-operatively (commencing from the arrival on the critical care unit, until the end of the 12th post-operative hour)
  To assess whether the presence of a central venous catheter influences the volume of intravenous fluid infused post-operatively

SECONDARY OUTCOMES:
Length of Intensive Care Unit Stay | From admission to intensive care, until stepdown to the ward (and until the expected end of study on 30th April 2020)
  Does the presence of a central venous catheter alter length of post-operative stay on the Intensive Care Unit
Volume of blood product infused peri-operatively | From induction of anaesthesia until the end of the 12th post-operative hour
  To assess whether the presence of a central venous catheter influences the volume of blood products infused peri-operatively
Mean dose of required vasopressor agents | From induction of anaesthesia until the end of the 12th post-operative hour
  To assess whether the presence of a central venous catheter influences the mean dose of any required vasopressor agents peri-operatively
Use of cardiac output (flow-monitoring) equipment | From induction of anaesthesia until the end of the 12th post-operative hour
  To assess whether the presence of a central venous catheter, and any ensuing fluid and blood pressure management strategies, influence the use of cardiac output monitoring equipment peri-operatively
Length of hospital stay | From the day of the procedure until discharge from the hospital (and until the expected end of study on 30th April 2020)
  To assess whether the presence of a central venous catheter influences the total post-operative length of stay

CONTACTS AND LOCATIONS:
Overall Officials: David Melia, MBBS, Study Director — Barts & The London NHS Trust
Locations (1):
- Whipps Cross Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At this stage there is no plan to make IPD available, and certainly no such intention has been discussed with the relevant ethical and review boards (HREC/HRA).